CLINICAL TRIAL: NCT04414540
Title: A Phase 2 Feasibility Study Combining Pembrolizumab and Metformin to Harness the Natural Killer Cytotoxic Response in Metastatic Head and Neck Cancer Patients
Brief Title: Combining Pembrolizumab and Metformin in Metastatic Head and Neck Cancer Patients
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Trisha Wise-Draper (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor-Investigator, Trisha Wise-Draper, Principal Investigator, University of Cincinnati
Organization: University of Cincinnati (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCCC-HN-19-01
Record Dates: First submitted 2020-05-11; First posted 2020-06-04 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Metformin; pembrolizumab

STUDY DESIGN:
Intervention Model Description: Patients will be on one of two arms that will be studied in parallel.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1: Metformin before Pembrolizumab (Experimental): Metformin ER 1000mg daily D-14 to D-7. Metformin ER 2000mg daily D-7 to D1. D1 Begin Pembrolizumab 200mg every 3 weeks, while continuing Metformin ER 2000mg daily.
  Interventions: Drug: Metformin Extended Release Oral Tablet; Drug: Pembrolizumab
- Arm 2: Metformin after Pembrolizumab (Experimental): D-21 Begin Pembrolizumab 200mg. D-7 begin Metformin ER 1000mg daily. D1 begin Metformin ER 2000mg daily. Continue Pembrolizumab 200mg every 3 weeks.
  Interventions: Drug: Metformin Extended Release Oral Tablet; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Metformin Extended Release Oral Tablet — Metformin ER starting dose 1000mg daily Metformin ER escalation dose 2000mg daily
  Other Names: Glucophage XR
Drug: Pembrolizumab — Pembrolizumab q 3 weeks
  Other Names: Keytruda

SUMMARY:
The purpose of this study is to determine anti-tumor activity by measuring overall response rate in recurrent and/or metastatic HNSCC patients receiving the combination of metformin and pembrolizumab.

DETAILED DESCRIPTION:
Recurrent and/or metastatic HNSCC patients will be treated with combination of metformin and pembrolizumab. Patients will be randomized into arms 1 and 2, to either receive Metformin prior to pembrolizumab or to begin Metformin after pembrolizumab treatment begins. The patients are randomized for the exploratory endpoints in order to better understand the difference of effects of metformin versus pembrolizumab on the immune system although efficacy is based on combination.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed recurrent or metastatic non-cutaneous HNSCC for which there are no surgical or radiation curative options.
* Patients may have received up to 3 prior lines of therapy for metastatic or recurrent disease.
* ECOG performance status ≤2

Exclusion Criteria:

* Patients with nasopharyngeal HNSCC will be excluded
* Patients who have had chemotherapy or radiotherapy within 2 weeks prior to entering the study.
* Patients who have not recovered from adverse events due to prior anti-cancer therapy
* Patients who have previously received PD-1 or PD-L1 inhibitors for metastatic/recurrent disease
* Patients currently receiving metformin or who have received metformin in the last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-08-31 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Overall Response by RECIST 1.1 and iRECIST | 2 years
  To determine anti-tumor activity by measuring overall response rate by RECIST 1.1 and iRECIST in recurrent and/or metastatic HNSCC patients receiving the combination of metformin and pembrolizumab.

SECONDARY OUTCOMES:
Number of patients with adverse events measured by CTCAE v5.0 | 2 years
  To observe and record safety of combination in metastatic HNSCC patients receiving the combination of metformin and pembrolizumab. AEs will be graded and recorded according to NCI CTCAE Version 5.0.
Progression Free Survival (PFS) | 1 year
  To observe and record progression free survival in recurrent and/or metastatic HNSCC patients receiving the combination of metformin and pembrolizumab.
Overall Survival (OS) | 1 year
  To observe and record overall survival in recurrent and/or metastatic HNSCC patients receiving the combination of metformin and pembrolizumab.

OTHER OUTCOMES:
Percentage of peripheral blood immune cell populations determined by flow cytometry | 4 weeks
  Peripheral blood will be collected from each treatment group
Percent tumor infiltrating NK cells determined by immunofluorescence | 4 weeks
  FFPE will be stained with NK cell antibodies to determine infiltrating NK cells
Cytokine levels including IL-2, IL-4, IL-6, IL-8, IL-10, INFgamma, TNFalpha in Plasma via ELISA based technology. | 4 weeks
  Plasma will be separated from peripheral blood from both treatment groups
Percentage of NK cell cytotoxicity via Natural Killer Cell Cytotoxicity Flow Based Assays. | 4 weeks
  Peripheral Blood separated for NK cells will be used from both treatment groups.
Stat-3 RNA levels in NK cells via RNA in situ | 4 weeks
  FFPE will be used from both treatment groups.
Percent secretion of NKG2D soluble ligands via ELISA. | 4 weeks
  Peripheral Blood will be used from both treatment groups

CONTACTS AND LOCATIONS:
Overall Officials: Trisha Wise-Draper, MD, PhD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No